CLINICAL TRIAL: NCT06435416
Title: Predictive Value of Postoperative Prognostic Nutritional Index Trajectory on 1-year Mortality After Off-pump Coronary Artery Bypass Surgery
Status: Completed | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Myung Il Bae, Clinical Assistant Professor, Gangnam Severance Hospital
Other Study IDs: 3-2023-0184
Record Dates: First submitted 2024-05-24; First posted 2024-05-30 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Patients Undergoing Off-pump Coronary Artery by Pass Surgery
Keywords: Prognostic Nutritional Index (PNI); Off-pump coronary artery bypass (OPCAB),; Coronary artery bypass graft surgery (CABG)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PNI trajectory group 1
  Interventions: Other: No intervention
- PNI trajectory group 2
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study investigated the changing pattern of postoperative Prognostic Nutritional Index (PNI) after off-pump coronary artery bypass surgery using a trajectory analysis. The investigators aimed to investigate the correlation between postoperative PNI recovery patterns and mortality in patients undergoing off-pump coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

• Patients aged ≥ 18 years who underwent off-pump coronary artery bypass surgery

Exclusion Criteria:

* Patients without PNI value between 1 and 3 days after surgery
* Patients without PNI value between 20 and 60 days after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing off-pump coronary artery bypass surgery
Sampling Method: Non-Probability Sample
Enrollment: 983 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
one-year mortality | one-year mortality after surgery
  1 year after surgery

SECONDARY OUTCOMES:
Overall mortality | Up to the last follow-up
  Overall mortality after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severnace Hospital, Seoul, GangnamGu, South Korea